CLINICAL TRIAL: NCT00209742
Title: Randomized Phase III Clinical Study Comparing Postoperative UFT+LV, UFT+LV/UFT and UFT+LV+PSK/UFT+PSK Therapies for Stage III Colorectal Cancer
Brief Title: Randomized Phase III Adjuvant Study for Stage III Colorectal Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hokkaido Gastrointestinal Cancer Study Group (Other)
Collaborators: Hokkaido University Hospital (Other)
Responsible Party: Yoshito Komatsu / A vice-director,, Hokkaido Gastrointestina Cancer Study Group
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HGCSG-CAD
Record Dates: First submitted 2005-09-12; First posted 2005-09-21 (Estimated); Last update posted 2010-05-26 (Estimated); Status verified 2010-05

CONDITIONS: Colorectal Cancer
Keywords: Colorectal Cancer,UFT,LV,Krestin,adjuvant therapy,phase III
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Tegafur; Leucovorin; polysaccharide-K

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 2 (Experimental)
  Interventions: Drug: UFT; Drug: USEL/Leucovorin
- 3 (Experimental)
  Interventions: Drug: UFT; Drug: USEL/Leucovorin; Drug: Krestin
- 1 (Active Comparator)
  Interventions: Drug: UFT; Drug: USEL/Leucovorin

INTERVENTIONS:
Drug: UFT — P.O. everyday
  Other Names: tegafur-uracil
Drug: USEL/Leucovorin — P.O. everyday
  Other Names: Leucovorin
Drug: Krestin — P.O. everyday
  Other Names: PSK
  Arms: 3

SUMMARY:
A randomized controlled study is conducted on patients with histological stage III colorectal cancer assigned to postoperative adjuvant therapy of uracil-tegafur plus leucovorin (UFT+LV), UFT+LV / UFT, or UFT+LV+PSK / UFT+PSK. The usefulness of the three regimens was evaluated by comparing the disease-free survival rate, overall survival rate, incidence and severity of adverse event, and quality of life.

DETAILED DESCRIPTION:
A multicenter randomized open-label controlled study is conducted on patients with histological stage III and curability A or B colorectal cancer [according to General Rules for Clinical and Pathological Studies on Cancer of the Colon, Rectum and Anus, 6th edition (Japanese Classification of Colorectal Cancer, English edition), also according to pTNM classification to facilitate overseas publication] given postoperative oral therapy of tegafur-uracil plus leucovorin (UFT+LV) (5 courses), UFT+LV (5 courses) / UFT (1 year), or UFT+LV+PSK (5 courses) / UFT+PSK (1 year). The usefulness of the three regimens as postoperative adjuvant therapy was evaluated by comparing the disease-free survival rate (DFR), overall survival rate (OS), incidence and severity of adverse event, and quality of life (QOL).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with primary colonic carcinoma or rectal carcinoma of histological stage III, who have undergone histological curability A or B surgeries
2. Patients evaluated histologically as lymph node metastasis positive
3. Patients aged between 20 and 80 years, inclusive, at the time of acquisition of informed consent
4. Patients with performance status 0 to 2
5. Patients who have not received preoperative cancer therapy (radiotherapy, chemotherapy or immunotherapy)
6. Gastrointestinal function: Patients with no diarrhea (watery stool)
7. Patients without severe impairment of renal, hepatic and bone marrow functions
8. Patients with no serious concurrent complications (such as infection)
9. Patients who have given written informed consent to participate in this study

Exclusion Criteria:

1. Patients graded as curability C
2. Patients with stenosis not capable of oral intake
3. Among disease stage IIIa cases, those that are si/n(-) and ai/n(-)
4. Patients with fresh hemorrhage from the gastrointestinal tract
5. Patients with retention of body fluid necessitating treatment
6. Patients with infection, intestinal palsy or intestinal occlusion
7. Patients with the lower end of the tumor involving the peritoneal reflection
8. Patients with lower rectal cancer (Rb), involving the anal canal (P) or perianal skin (E)
9. Patients with active multiple cancers; or even if the multiple cancers are metachronous, have a disease-free period of less than 5 years (but excluding cancer in situ and skin cancer)
10. Patients who are pregnant or hope to become pregnant during the study period
11. Patients with poorly controlled diabetes or are treated by continuous use of insulin
12. Patients with a history of ischemic heart disease
13. Patients with concurrent psychiatric disease or psychotic symptoms, and judged to have difficulties participating in the study
14. Patients receiving continuous administration of steroids
15. Patients who have experienced serious drug allergy in the past
16. Others, patients judged by the investigator or subinvestigator to be inappropriate as subject

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Estimated)
Dates: Start 2005-04; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
3-years disease-free survival rate (DFS) | 5-years

SECONDARY OUTCOMES:
Dose intensity (compliance), 5-year disease-free survival rate, 3- and 5-year survival rate, incidence of other adverse drug reactions, QOL | 7-years

CONTACTS AND LOCATIONS:
Overall Officials: Masahiro Asaka, MD, PhD, Study Chair — Hokkaido Gastrointestinal Cancer Study Group
Locations (1):
- ・ Hokkaido University Hospital (Hokkaido University Graduate School of Medicine / School of Medicine), Sapporo, Hokkaido, Japan